CLINICAL TRIAL: NCT03933176
Title: Is the Use of a Glass Ionomer Liner Necessary After Selective Carious Tissue Removal?
Brief Title: Absence of Liner Following the Selective Caries Removal (ALFSCaRe)
Acronym: (ALFSCaRe)
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: COVID-19 pandemic
Sponsor: Universidade Federal de Sergipe (Other)
Collaborators: Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government); Federal University of Pelotas (Other); University of Brasilia (Other); Universidade Federal do Ceara (Other); Federal University of Uberlandia (Other); Universidade Veiga de Almeida (Other)
Responsible Party: Principal Investigator, André Luis Faria e Silva, Professor, Universidade Federal de Sergipe
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UFS/Prodonto
Record Dates: First submitted 2019-04-26; First posted 2019-05-01 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Caries; Dentin; Dental Restoration Failure of Marginal Integrity
Keywords: Glass ionomer; Bulk-Fill Composite

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Simplified restorative procedure (Experimental): After selective carious tissue removal, the universal adhesive (Adper Universal; 3M ESPE, St. Paul, MN, EUA) will be applied on the cavity walls. The cavity will be restored using a single increment of Filtek One Bulk Fill (3M ESPE, St. Paul, MN, EUA).
  Interventions: Procedure: Restoration of carious lesions
- Control (Active Comparator): A thin layer of resin-modified glass ionomer (Ionoseal (Voco America Inc., Briarcliff Manor, NY, EUA) will be placed on the pulpal floor of the cavity. Then, the adhesive and composite will be used following the same directions defined for the experimental condition.
  Interventions: Procedure: Restoration of carious lesions

INTERVENTIONS:
Procedure: Restoration of carious lesions — Selective carious tissue removal followed by restoration of the cavity using composite resin.

SUMMARY:
This randomized, multi-centric, controlled clinical trial will assess the effectiveness of a simplified restorative protocol used after the selective carious tissue removal in posterior teeth presenting deep carious lesions. Only a regular bulk-fill composite will be used in the simplified restorative protocol following the application of universal adhesive. A liner with resin-modified glass ionomer will be used over the pulpal floor before the composite placement in the control group. The longevity of restorative procedures and post-operative sensitivity were defined as the main and secondary outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Molar presenting deep carious lesion;

Exclusion Criteria:

* Non-vital teeth or teeth presenting pulpitis;
* Cavity margins in dentin;
* Presence of non-carious cervical lesions;
* The necessity of restoration involving any cusp replacement.

Ages: 6 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2019-06-30 (Actual); Primary Completion 2020-11-01 (Actual); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Longevity of restoration | Annual evaluation during 5 years
  Assessment of any failure in restorations according to the FDI World Dental Federation criteria.

SECONDARY OUTCOMES:
Tooth sensitivity | 15 days after the restorative procedure
  The participants will self-assess their level of tooth sensitivity of the restored teeth using a visual analogue scale of 0-10 (0 indicating absence of pain; and 10 the worst pain possible) oriented by both verbal description and Wong-Baker facial grimace scales.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Dentistry/ Federal University of Sergipe, Aracaju, Sergipe, Brazil

IPD SHARING:
Plan to Share IPD: Undecided